CLINICAL TRIAL: NCT01552577
Title: Eye Tracking Indicators of Neurocognitive Status After Traumatic Brain Injury
Brief Title: The RETINA Project: Reliable Eye Tracking in Neurocognitive Assessment of Traumatic Brain Injury
Acronym: RETINA
Status: Terminated | Type: Observational
Why Stopped: Expiration of funding
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mark Ettenhofer, Assistant Professor, Uniformed Services University of the Health Sciences
Other Study IDs: R072LP-SS3
Record Dates: First submitted 2012-03-08; First posted 2012-03-13 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Traumatic Brain Injury
Keywords: Post-Concussion Syndrome; Concussion; Brain Injury; TBI; Military Personnel; Eye-tracking; Neurocognitive Function; Assessment
MeSH Terms: conditions — Brain Injuries, Traumatic; Post-Concussion Syndrome; Brain Concussion; Brain Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- TBI Group: Adults (civilian or military) with a history of one or more brain injuries / concussions.
- Control Group: Healthy adults (civilian or military) with no history of brain injury.

SUMMARY:
The purpose of this study is to develop and validate eye-tracking measures that can be used to evaluate neurocognitive dysfunction among individuals with traumatic brain injury (TBI).

DETAILED DESCRIPTION:
This study will evaluate a novel method of neurocognitive assessment using computerized eye tracking. This method involves looking at targets on a computer screen while an eye-tracking system records eye movements and changes in pupil diameter in response to the presentation of the targets.

Performance on the eye tracking measures will be evaluated to identify potential effects of neural injury on cognitive performance. Data from individuals with and without a history of brain injury will be used to standardize the eye tracking measure.

Participants will also complete a short interview and several self report measures, including information about demographic characteristics, medical history, and psychological symptoms, along with a series of neuropsychological/cognitive measures that are already well established. Performance on eye tracking measures will then be compared to performance on these conventional cognitive tests to allow comparison of the different measures.

All participants will complete one visit to the laboratory at USUHS in Bethesda, MD. This visit will take approximately 2.5 hours. Participants without a history of TBI may be asked to return for a 30 minute follow-up session in order to measure the reliability of the eye tracking system. Participants with a history of TBI will complete a 10 minute telephone follow-up 6 and 12 months after their visit.

Compensation is available for civilians who are not employed by the Federal government.

ELIGIBILITY:
Inclusion Criteria (Control Group):

* 18 years of age or older
* No history of brain injury or concussion
* Fluency and literacy in English
* Can effectively communicate verbally
* Willing and able to provide written informed consent
* Obtains signed permission to participate from supervisor and/or brigade commander (federal civilian employees and active duty military personnel only).

Exclusion Criteria (Control Group)

* Impaired or fluctuating level of consciousness / arousal
* Any medical condition that could impair cognitive abilities (e.g. muscular dystrophy, multiple sclerosis, psychosis)
* History of any neurological conditions such as brain tumor, brain infection, seizure or stroke
* Any visual impairment that is not corrected by glasses/contacts
* Motor impairment or amputation of one or both upper extremities

Inclusion Criteria (TBI Group):

* 18 years of age or older
* History of one or more brain injuries / concussion
* Fluency and literacy in English
* Can effectively communicate verbally
* Willing and able to provide written informed consent
* Obtains signed permission to participate from supervisor and/or brigade commander (federal civilian employees and active duty military personnel only).

Exclusion Criteria (TBI Group)

* Impaired or fluctuating level of consciousness / arousal
* Any medical condition that could impair cognitive abilities (e.g. muscular dystrophy, multiple sclerosis, psychosis), other than TBI
* History of any neurological conditions (such as brain tumor, brain infection, seizure or stroke) that was NOT associated with or resulting from traumatic brain injury
* Any visual impairment that is not corrected by glasses/contacts
* Motor impairment or amputation of one or both upper extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population to be studied will include civilians and military personnel with and without a history of traumatic brain injury / concussion.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2010-10; Primary Completion 2015-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Performance on the eye tracking measures | Baseline

SECONDARY OUTCOMES:
Psychological symptoms | Baseline
Performance on the neurocognitive assessment battery | Baseline
Post-concussive symptoms | Baseline (and telephone follow-up, for TBI group)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ettenhofer, Ph.D, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- USUHS, Bethesda, Maryland, United States